CLINICAL TRIAL: NCT01507883
Title: Time-lapse Evaluation of Human Embryo Development in Single Versus Sequential Culture Media - a Sibling Oocyte Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bahceci Health Group (Other)
Responsible Party: Principal Investigator, H. NADIR CIRAY, Associate Professor, MD., PhD, Bahceci Health Group
Other Study IDs: BHC1
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: In-vitro Fertilization
Keywords: Supervision; embryos; Resulting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human embryos
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- human oocytes/embryos: Sibling oocytes cultured in single or sequential media until day6

SUMMARY:
Current human IVF technology employs two strategies with respective culture media for embryo development; 'let the embryo choose' (utilizes single step media) and 'back-to-nature' (utilizes sequential media). To our knowledge, there is not any sibling oocyte study to evaluate potential advantages/disadvantages of these strategies on one another.

DETAILED DESCRIPTION:
Maintaining optimal embryo development during in vitro culture is a key element in assisted reproduction treatments. Whether the concept of mimicking in vivo environment is a 'must' in order not to compromise outcome is a matter of debate since 'let the embryo choose' strategy has been shown to perform at least as good as the 'back to nature' in several studies.'Let the embryo choose" approach utilizes a milieu with relatively constant concentration of ingredients (single culture system) as compared to the latter, in which demands of the embryos are supported according to their passage from the Fallopian tubes to the uterus in a sequential culture media. Basic differences between these ingredients are; presence of (1) glucose instead of pyruvate, and (2) essential aminoacids in early embryo stages (until day 3) in single step media, and (3) presence of EDTA in sequential media.

Vast majority of these results were obtained from studies where patients have been randomized into groups instead of employing a sibling (oocyte/embryo) model which could have enabled each patient to serve as her own control. In fact, it has been claimed that introducing a sibling oocyte study design could give a methodological problem at the time of fertilization since different type of culture media vary in osmolarity. Likewise the only study that employed a sibling oocyte model utilized two different media (home-made versus G1.2/G1.2) although the osmolarity of the former had been adjusted to 280-285 mOsm). This study reported no significant differences in day3/5 embryo development as well as pregnancy/implantation rates between groups.

Subsequent studies, however, favoured single step media, as they found higher proportion of compacted embryos to zygotes at day3, morula at 4, a higher blastocyst yield, an overall higher utilization rate after day5 and an improved implantation rate when compared to sequential media. Yet, besides potential variation of gamete qualities between patients allocated to groups (as described above), differences in static observation times of embryos between laboratories could have affected the results in these studies. Current introduction of time-lapse equipment into human assisted reproduction technology enabled a more distinct definition of embryo development and it is now possible to quantify pace of embryo cleavage in various media. Such a definition is also useful to determine the predictive value of embryo development in pre-defined time points will be applicable to all embryology laboratories using various culture systems.

ELIGIBILITY:
Inclusion Criteria:

* Cycles which have gone through egg retrieval procedure between March to November 2011 were included into the study.There was no restriction on the number of previous trials and/or sperm source.

Exclusion Criteria:

* The maximum number of retrieved oocytes was restricted to 12 and the minimum to 2, as the former was the capacity of one dish (EmbryoSlide™) in which oocytes/embryos could be placed and the latter was the minimum number to be able to make a comparison between groups. Women who were older than 40 years of age were excluded in order to minimize the impact of increased risk of aneuploidy on the results.
* Cycles in which oocytes/embryos have been subjected to biopsy were also excluded due to the potential risk of delayed embryo development in such cases (Kirkegaard et al., 2011).
* Furthermore, cycles in which diagnosis of infertility was endometrial factor were not included since such aetiology could negatively affect implantation despite good embryo development.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who had undergone infertility treatment and oocytes subjected to ICSI
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nadir H Ciray, MD., PhD, Principal Investigator — Bahceci Health Group; Turan Aksoy, BS, Study Chair — Bahceci Health Group; Mustafa Bahceci, MD, Study Director — Bahceci Health Group; Cihan Goktas, BS, Study Chair — Bahceci Health Group; Birgen Ozturk, BS, Study Chair — Bahceci Health Group
Locations (1):
- Bahceci Fulya IVF Clinic, Istanbul, Turkey (Türkiye)